CLINICAL TRIAL: NCT06553014
Title: Effectiveness of Endovascular Plug Embolization in Pelvic Congestion Syndrome
Status: Completed | Type: Observational
Sponsor: Halil Ibrahim Altun (Other)
Responsible Party: Sponsor-Investigator, Halil Ibrahim Altun, pain specialist, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: ibrahim
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pain, Chronic
Keywords: Pelvic Congestion Syndrome, Pain,chronic pelvic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Effectiveness of Endovascular Plug Embolization in Pelvic Congestion Syndrome: Effectiveness of Endovascular Plug Embolization in Pelvic Congestion Syndrome
  Interventions: Other: Endovascular Plug Embolization

INTERVENTIONS:
Other: Endovascular Plug Embolization — Effectiveness of Endovascular Plug Embolization in Pelvic Congestion Syndrome

SUMMARY:
Pelvic Congestion Syndrome (PKS) is generally seen in female patients of reproductive age and is characterized by abdominopelvic pain and a feeling of fullness in the perineum and vulva. Patients may also be accompanied by dysmenorrhea , dyspareunia, postcoital pain, dysuria , hematuria, waist and hip pain. The pain usually increases with standing and decreases with lying down. PCS is one of the causes of chronic pelvic pain (CPA). As in CPA , it lasts longer than 6 months and is independent of the menstrual cycle. Its etiopathogenesis has not been fully elucidated. at PKS There is dilatation in the ovarian veins. In the current definition, diseases that involve dilatation of the veins in the pelvic region and were referred to by different names in the past are called Pelvic Venous Disease .

There is no consensus on the diagnostic criteria for PCS . Catheter venography along with the patient's clinical findings is still the gold standard in diagnosis. Among non- invasive methods , >0.6 mm dilatation in the ovarian veins on transvaginal or transabdominal ultrasound (USG) is one of the most important findings of PCS .

There have been significant changes in its treatment in recent years. Some of the hormone treatments used in the 1980s were abandoned due to their side effects. Some flavonoid fraction drugs are used in PCS due to their vasoactive effects . Anti-inflammatory drugs, paracetamol, are preferred for analgesic purposes , and gabapentinoids and antidepressants are preferred for central sensitization . In the same years, hysterectomy and single or bilateral oophorectomy were performed by gynecologists. Laparoscopic ovarian vein ligation began to be performed in the 2000s , but it lost its popularity due to serious complications such as hematoma in the retroperitoneum and ureteral injury . Today, some endovascular sclerosing drugs, foam, plug and coil embolization techniques are frequently used alone or in combination in the treatment of PCS . There are studies on the low complications and high effectiveness of these treatments .

Diagnosis and treatment of PCS patients, who frequently apply to urology and gynecology, are often delayed, patients are followed up with different diagnoses, and the cost increases. Endovascular intervention is a minimally invasive technique and patients are discharged on the same day. There are approximately 3 times more studies in the literature ( PUBMED, EMBASE, MEDLINE (OVID), Web of Science ) on coil embolization , one of the endovascular methods used , than on plug treatment (9). We aimed to contribute to the limited literature on the effectiveness of plug therapy in PCS patients with limited access to diagnosis and treatment .

DETAILED DESCRIPTION:
Patients diagnosed with pelvic congestion syndrome who underwent endovascular procedures using the plug method in the cardiovascular surgery clinic of our hospital between January 2023 and March 2024 were examined. The study was conducted in accordance with the Declaration of Helsinki. The study was conducted retrospectively with 32 patients who met the criteria.

18 years of age , with abdominopelvic pain for more than 6 months , with clinical, physical examination and symptoms , and with >6 mm dilatation in the pelvic veins on transvaginal or transabdominal ultrasound (USG) were included in the study. It was performed by a radiologist with at least 10 years of experience in the field of USG.

Gynecologically, patients with leiomyoma, pelvic inflammatory disease, endometriosis , postoperative adhesion, patients who have undergone urological and gynecological surgery, patients with chronic renal failure, patients with known allergies to the drugs used during the procedure , patients with abdominopelvic trauma, malignancy or its history, patients with a history of radiotherapy chemotherapy, patients with known psychiatric disease, Pregnant women, breastfeeding women, patients with fibromyalgia , known lumbar disc herniation, scoliosis, facet syndrome, sacroiliac dysfunction, and patients with genitourinary and gastrointestinal diseases were excluded from the study.

Patients' age, body mass index (BMI), painful areas (perineum, vulva, labia major/minor, hypogastrium , inguinal region, hip, waist, leg) and painful side, medical treatments, additional diseases, onset of pain and application for endovascular intervention. duration, symptoms accompanying pain ( feeling of heaviness in the perineum , labia swelling in the majora , Dysuria , Hematuria, Dyspareunia , Postcoital pain, Dysmenorrhea , frequent urination) In which position does the pain increase: lying down: (supine / prone / lateral) standing / sitting, presence of varicose veins in the lower extremity , vein entered during endovascular intervention, embolized vein, embolotherapy type, procedure time (min), cumulative radiation exposure during the procedure (mGy- m2 ) Complications observed during the procedure (Vessel perforation / Hematoma / Phlebitis / Embolism / Migration / Vasovagal / Dyspnea / Panic attack / Allergy / Infection) and the need for repeated procedures were recorded in the patient follow-up form.

For pain and functionality evaluation, NRS-11 scores and SF-12 scores were recorded before and at the first and third months after the endovascular procedure.

1. Numeric Rating Scale-11 ( NRS - 11 ) is an 11-point numerical scale where patients can evaluate their pain between 0 (no pain) and 10 (the most severe pain they have ever felt in their life) .
2. Short form-12 (SF-12): It is a scale that evaluates patients' quality of life levels. Short Form-12 is the abbreviation of Short Form-36. In SF-12, the patient's general health status, physical and mental functions, quality of life and social activities are questioned. It is scored between 0-100. A high score is associated with good general health status. It is a validated scale. This test was applied 3 times: before treatment, 1 month and 3 months after treatment.

ELIGIBILITY:
exclusion criteria: -Gynecologically, patients with leiomyoma, pelvic inflammatory disease, endometriosis , postoperative adhesion,

* Patients who have undergone urological and gynecological surgery,
* Patients with chronic renal failure,
* Patients with known allergies to the drugs used during the procedure ,
* Patients with abdominopelvic trauma, malignancy or its history,
* Patients with a history of radiotherapy chemotherapy,
* Patients with known psychiatric disease,
* Pregnant women,
* Breastfeeding women,
* Patients with fibromyalgia ,
* Known lumbar disc herniation, scoliosis, facet syndrome, sacroiliac dysfunction, and patients with genitourinary and gastrointestinal diseases were excluded from the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * 18 years of age
  * with abdominopelvic pain for more than 6 months ,
  * with clinical, physical examination and symptoms , and with >6 mm dilatation in the pelvic veins on transvaginal or transabdominal ultrasound (USG) were included in the study.
  * It was performed by a radiologist with at least 10 years of experience in the field of USG
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
onset of pain and application time for endovascular intervention | 'four months'

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)